CLINICAL TRIAL: NCT00369642
Title: A Controlled Trial of Daily Cognitive-Behavioral Therapy for Pediatric Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF212-2004
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2008-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Cognitive-behavioral therapy; Children; Obsessive-compulsive disorder; Intensive Cognitive-behavioral therapy; Weekly Cognitive-behavioral therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy

SUMMARY:
Pediatric obsessive-compulsive disorder (OCD) is a chronic and often disabling illness with an estimated lifetime prevalence of 1 to 3%. Pediatric OCD is associated with significant social, educational, and familial impairment, as well as comorbid emotional and behavioral disturbances that serve to complicate the prognosis of the illness and treatment outcome. While limited open treatment trials and one controlled trial have demonstrated cognitive-behavioral therapy (CBT) to be effective for pediatric OCD, controlled trials are lacking in the literature. There are a number of incremental benefits that an intensive program for OCD may offer. First, existing outpatient interventions typically achieve treatment gains over a 15 to 20 week period. The present program typically lasts between 2 to 4 weeks, and thus may present as a more timely, cost-effective, and efficient means of treatment for some individuals. Second, given that many children and adolescents may not have access to mental health professionals who are trained in empirically grounded interventions for OCD, the present treatment setting allows youth to receive appropriate, state of the art care. Finally, evidence suggests that daily CBT may be particularly effective in treating children who have been refractory to prior treatments (e.g., medication or once per week CBT). Prior to treatment, all consenting families will be randomly assigned to either the treatment condition or a three-week wait-list control condition. Those families randomized to the wait-list condition will receive treatment immediately after the three weeks are completed. The treatment group will be administered all measures immediately before treatment, immediately after treatment, and three months after treatment. The wait-list control condition will be administered all measures upon starting the wait-list period, immediately following the conclusion of the three-week wait-list period, and after the treatment program has finished. The purpose of the current study is to evaluate the efficacy of daily cognitive-behavioral treatment for pediatric OCD.

DETAILED DESCRIPTION:
Distressing, intrusive thoughts, images, or impulses and repetitive mental or behavioral rituals aimed to reduce distress are the hallmark of adult and pediatric obsessive-compulsive disorder (OCD). Epidemiological studies suggest a prevalence rate of between 1 to 4% in children and adolescents (Douglass, Moffitt, Dar, McGee, & Silva, 1995; Flament, Whitaker, Rapoport, & Davies, 1988; Zohar, 1999). If untreated, OCD is related to significant social, academic, and familial impairment (Koran, Thienemann, & Davenport, 1996; Piacentini et al., 2003).

Cognitive-behavioral therapy (CBT) is a form of psychotherapy with proven efficacy for OCD treatment in adult populations (see Franklin & Foa, 2002 for a review). More recently, several open (Benazon, Ager, & Rosenberg, 2002; March, Mulle, & Herbel, 1994; Piacentini, Bergman, Jacobs, McCracken, & Kretchman, 2002) and one controlled trial (de Haan, Hoogduin, Buitelaar, & Keijsers, 1998) have supported the effectiveness of this approach with children and adolescents diagnosed with OCD. Cognitive-behavioral therapy for adult and pediatric OCD can be broken down into two general components. First, in exposure and response prevention (ERP), patients are gradually exposed to anxiety-provoking stimuli while refraining from engaging in compulsive behaviors or rituals (Meyer, 1966). The extended exposure to anxiety-provoking stimuli causes anxiety to habituate and provides objective data that contradicts inaccurate expectations of harm and responsibility (Foa & Kozac, 1996). Second, cognitive therapy teaches the patient to identify and correct anxiety-provoking cognitions that often motivate compulsive behaviors. Objective, realistic cognitions that are not linked to obsessive-compulsive anxiety will result in reduced needs to perform compulsive acts.

Although the results of the above mentioned psychotherapy trials, as well as a number of pharmacological treatment trials, are promising (Cook et al., 2001; DeVeaugh-Geiss, Moroz, Biederman, & Cantwell, 1992; Geller et al., 2001; Liebowitz et al., 2002; March et al., 1998; Riddle et al., 2001), it is important to note that a relatively large number of patients do not respond to treatment in a clinically significant manner. For example, the treatment response rates in recent major drug trials ranged from 42 to 67% (Cook et al., 2001; DeVeaugh-Geiss et al., 1992; Geller et al., 2001; Liebowitz et al., 2002; Riddle et al., 2001), whereas the treatment response rate in the referenced psychotherapy trials ranged from 63 to 79%. As such, it is important to identify and test potential treatment approaches that may be suitable for treatment refractory pediatric OCD patients.

One manner of treating children with OCD who do no adequately respond to conventional medication or psychotherapy interventions is through intensive CBT. The UF OCD Program in the Department of Psychiatry at the University of Florida utilizes the principles of CBT. Our intensive program provides CBT services to children on an outpatient basis. Intensive outpatient treatment involves the child and his/her parent(s) or guardian(s) moving to Gainesville for three weeks, which usually requires staying in a hotel, unless the person has friends or relatives living in the area. Patients are seen five days per week for approximately three weeks. Sessions typically involve exposure and response prevention in conjunction with cognitive therapy for older children. Family members are involved extensively in treatment to assist with the completion of daily homework exercises and generalization of skills to the home environment. In addition to being an alternative approach for treatment refractory youth, there are a number of other benefits that an intensive program for pediatric OCD may offer. First, an intensive approach may be well suited for children with severe symptomatology or functional impairment (e.g., not going to school; Franklin, Tolin, March, & Foa, 2001; Storch, Gelfand, Geffken, & Goodman, 2003). Second, existing outpatient interventions typically achieve treatment gains over a 15 to 20 week period. Intensive treatment typically lasts three to four weeks, and thus may present as a more timely, cost-effective, and efficient means of treatment, particularly when the child is missing out on important normative events (e.g., school attendance). Third, many people do not have access to mental health professionals who are trained in empirically grounded OCD treatment and thus, are unable to receive the most effective care. For example, Flament et al. (1988) found that only 22% of a sample of children with OCD were receiving mental health services. Moreover, none of those being treated were receiving appropriate, empirically validated intervention. Finally, time-limited, intensive programs may enhance the child's motivation by becoming the primary focus for several weeks, which may not be the case with standard weekly treatment (Foa & Steketee, 1987).

Although several open and controlled trials of intensive psychotherapy for adult OCD have been published (Abramowitz, Foa, & Franklin, 2003; Cottraux et al., 2001; Foa, Kozak, Steketee, & McCarthy, 1992; Storch et al., 2003), to date, only two examples of intensive outpatient treatment for OCD in childhood has been reported (Franklin et al., 2001; Storch et al., 2004). Franklin et al. (2001) describes a 12-year-old boy with severe OCD who was seen five days per week for a total of 11 sessions. Results indicated marked improvements in clinician-rated OCD symptoms and self-reported depressive symptoms. Storch et al. (2004) provides data on five children with OCD consecutively seen in intensive cognitive-behavioral psychotherapy. Assessments were conducted at baseline and after treatment. All participants were classified as treatment responders (much improved or very much improved). Two of the participants did not meet diagnostic criteria for OCD following treatment. The severity of clinician-rated OCD symptoms and impairment significantly decreased after the intervention.

Under the proposed controlled trial, we plan to examine the efficacy of daily cognitive-behavioral psychotherapy to 50 consecutive children and adolescents who enroll in the UF OCD program. Children will be randomized to one of two treatment conditions: one consists of receiving cognitive-behavioral therapy every weekday for three-weeks; the other consists of receiving treatment as usual, which consists of once per week outpatient cognitive-behavioral therapy sessions . As compared to the once per week therapy condition, we predict decreases in OCD, general anxiety, and depressive symptomatology, and functional impairment at post-intervention for youth in the daily therapy condition.

ELIGIBILITY:
Inclusion Criteria:

1. CY-BOCS Total Score ≥ 16;
2. no change in psychotropic medication (if applicable) for at least 8 weeks prior to study entry;
3. 7 to 17 years old; and
4. availability of at least one parent to accompany the child to all treatment sessions.

Exclusion Criteria:

1. history of and/or current psychosis, pervasive developmental disorder, bipolar disorder, or current suicidality measured by the ADIS-IV-P and all available clinical information;
2. principal diagnosis other than OCD;
3. a positive diagnosis in the caregiver of mental retardation, psychosis, or other psychiatric disorders or conditions that would limit their ability to understand CBT (based on clinical interview). Participants were not excluded due to comorbid psychiatric diagnoses.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2004-10; Study Completion 2006-12

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS; Scahill et al., 1997)
Clinical Global Impression - Severity (CGI-S; National Institute of Mental Health, 1985)
Clinical Global Improvement (CGI; Guy, 1976)

SECONDARY OUTCOMES:
Multidemisional Anxiety Scale for Children
Children's Depression Inventory
Family Accommodation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Pediatric OCD Treatment Study (POTS) Team. Cognitive-behavior therapy, sertraline, and their combination for children and adolescents with obsessive-compulsive disorder: the Pediatric OCD Treatment Study (POTS) randomized controlled trial. JAMA. 2004 Oct 27;292(16):1969-76. doi: 10.1001/jama.292.16.1969. PMID 15507582
- [Derived] Storch EA, Merlo LJ, Larson MJ, Geffken GR, Lehmkuhl HD, Jacob ML, Murphy TK, Goodman WK. Impact of comorbidity on cognitive-behavioral therapy response in pediatric obsessive-compulsive disorder. J Am Acad Child Adolesc Psychiatry. 2008 May;47(5):583-592. doi: 10.1097/CHI.0b013e31816774b1. PMID 18356759